CLINICAL TRIAL: NCT06327321
Title: Vitiligo Treatment by Targeting TYK2 Mediated Responses Prospective Multicentric Double Blind Interventional Study
Brief Title: Vitiligo Treatment by Targeting TYK2 Mediated Responses
Acronym: ViTYK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23-PP-08
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Vitiligo, Generalized
MeSH Terms: conditions — Vitiligo | interventions — deucravacitinib; Therapeutics

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug group (Experimental): Following central randomization, patients will be assigned to receive either deucravacitinib 12mg daily (QD) or a placebo daily (QD) for a duration of 24 weeks. At the end of this period, patients will be re-randomized to receive either deucravacitinib 12mg QD alone or deucravacitinib 12mg QD + twice weekly narrowband UVB treatment twice weekly for an additional 24 weeks.
  Interventions: Drug: Deucravacitinib
- Placebo group (Placebo Comparator): Following central randomization, patients will be assigned to receive either deucravacitinib 12mg daily (QD) or a placebo daily (QD) for a duration of 24 weeks. At the end of this period, patients will be re-randomized to receive either deucravacitinib 12mg QD alone or deucravacitinib 12mg QD + twice weekly narrowband UVB treatment twice weekly for an additional 24 weeks.
  Interventions: Other: Volunteer without treatment

INTERVENTIONS:
Drug: Deucravacitinib — Throughout the study, there will be a total of six visits conducted: selection, inclusion, Week 12, Week 24, Week 36, and Week 48. In patients who volunteer, a skin biopsy will be performed on both the lesional and peri-lesional areas at baseline, Week 12 and Week 36. Serum and plasma samples will be collected at the screening visit, Week 12, Week 24, Week 36, and Week 48.
  Arms: Drug group
Other: Volunteer without treatment — Throughout the study, there will be a total of six visits conducted: selection, inclusion, Week 12, Week 24, Week 36, and Week 48. In patients who volunteer, a skin biopsy will be performed on both the lesional and peri-lesional areas at baseline, Week 12 and Week 36. Serum and plasma samples will be collected at the screening visit, Week 12, Week 24, Week 36, and Week 48.
  Arms: Placebo group

SUMMARY:
Vitiligo affects approximately 1 to 2% of the global population and significantly impacts people's quality of life. Achieving the best treatment outcomes for vitiligo involves addressing the autoimmune inflammatory response to stop the depigmentation process and promoting the differentiation of melanocyte stem cells to induce repigmentation. The loss of melanocytes in vitiligo is a result of an autoimmune process. While the IFN gamma pathway plays a crucial role in the adaptive immune response in vitiligo, there is increasing evidence highlighting the importance of the innate immune response. Deucravacitinib, an allosteric TYK2 inhibitor, has shown effectiveness and safety in treating psoriasis. It inhibits the responses of IFN alpha (IFNα), IFN beta (IFNβ), and IL12, and may also have an impact on the Th1 response. The hypothesis is that by targeting the IFN type I response and IL12, deucravacitinib could effectively halt the depigmentation process and facilitate repigmentation of vitiligo lesions. When combined with NB-UVB, the process of repigmentation should be significantly enhanced. The primary objective is to compare the proportion of patients treated with deucravacitinib versus placebo achieving VITIL-IA 50 at week 24.

Interventions Following central randomization, patients will be assigned to receive either deucravacitinib 12mg daily (QD) or a placebo daily (QD) for a duration of 24 weeks. At the end of this period, patients will be re-randomized to receive either deucravacitinib 12mg QD alone or deucravacitinib 12mg QD + twice weekly narrowband UVB treatment twice weekly for an additional 24 weeks.

Throughout the study, there will be a total of six visits conducted: selection, inclusion, Week 12, Week 24, Week 36, and Week 48. In patients who volunteer, a skin biopsy will be performed on both the lesional and peri-lesional areas at baseline, Week 12 and Week 36. Serum and plasma samples will be collected at the screening visit, Week 12, Week 24, Week 36, and Week 48.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women with non-segmental vitiligo.
2. ≥ 18 and <75 years
3. Patient with at least one lesion of more than 2 cm² not located on the face, hands or feet.
4. Patients with Vitil-IA score above 5% and T-VASI above 5% (not taking into account the involvement of hands and feet)
5. For women of child-bearing age, an effective contraception (estroprogestative pill, contraceptive implant, IUD, condoms or tubal ligation) should be used for more than one month before the inclusion in the study. A urine pregnancy test (βHCG in urines) will be performed.
6. Affiliation to a social security system
7. Signed informed consent
8. Patient willing and able to attend all study visits

Exclusion Criteria:

1. Pregnant or breast-feeding women. Or women with potential childbearing and not taking contraceptives or who plan to get pregnant during the study duration.
2. Segmental or mixed vitiligo
3. Concomitant use of topical or systemic immunosuppressive medication or steroids
4. Patients suffering from photodermatosis or taking photosensitive drugs
5. Personal history of skin cancer
6. Personal history of cancer of less than 5 years
7. Patients with active infection
8. Tuberculosis or latent tuberculosis
9. Vulnerable people: pregnant or breast-feeding women, minors, adult under guardianship or deprived of freedom
10. Participants in other clinical therapeutic studies involving a drug that could interfere with the present evaluation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2026-05-05 (Estimated); Study Completion 2026-11-05 (Estimated)

PRIMARY OUTCOMES:
rate of depigmentation | at week 24
  Improvement of at least 50% of the depigmentation of the face assessed by the Vitil-IA algorithm on UV pictures performed on ColorFace (Vitil-IA 50)

SECONDARY OUTCOMES:
number of patient with the T-VASI 50 | at 48 weeks

CONTACTS AND LOCATIONS:
Overall Officials: PASSERON Thierry, PhD, Principal Investigator — CHU de Nice, Service de Dermatologie
Locations (5):
- France (5):
  - CHU de Nice - Hôpital de l'Archet, Nice, Alpes-Maritimes
  - APHP, Henri Mondor, Paris, Creteil
  - CHU de Bordeaux, Bordeaux, Talence
  - CHU de Lille, Lille
  - HCL, Lyon